CLINICAL TRIAL: NCT06873711
Title: The Associations of Microribonucleic Acid Gene Polymorphisms With the Risk and Clinicopathological Characteristics of Ulcerative Colitis
Brief Title: The Associations of Microribonucleic Acid Gene Polymorphisms With the Risk of Ulcerative Colitis
Status: Completed | Type: Observational
Sponsor: Second Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: SAHoWMU-CR2025-01-206
Record Dates: First submitted 2025-03-02; First posted 2025-03-13 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Colitis, Ulcerative
MeSH Terms: conditions — Colitis, Ulcerative | interventions — vedolizumab

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Extract whole genome DNA from peripheral blood
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- UC patients: Some UC patients received intravenous injection of VDZ (300mg/time) at weeks 0, 2, and 6, followed by intravenous injection of the same dose of VDZ every 8 weeks to maintain treatment.
  Interventions: Biological: vedolizumab
- normal control: no biological agents treatment

INTERVENTIONS:
Biological: vedolizumab — Intravenous injection of VDZ (300mg/time) at weeks 0, 2, and 6, followed by intravenous injection of the same dose of VDZ every 8 weeks to maintain treatment.
  Groups: UC patients

SUMMARY:
From January 2020 to December 2024, diagnosed ulcerative colitis(UC) patients and gender- and age-matched normal controls were enrolled from the Department of Gastroenterology, the Second Affiliated Hospital of Wenzhou Medical University. Our aim is to investigate the associations of microribonucleic acid(miRNA) gene polymorphisms with the risk and clinicopathological characteristics of UC, and to analyze the effects of miRNAs gene variations on the clinical response of vedolizumab(VDZ) treatment in UC patients.

DETAILED DESCRIPTION:
From January 2020 to December 2024, diagnosed UC patients and gender- and age-matched normal controls were enrolled from the Department of Gastroenterology, the Second Affiliated Hospital of Wenzhou Medical University. Genotypes of miRNAs were determined by multiplex polymerase chain reaction-ligase detection reaction technique. Chi-square test and unconditional logistic regression model were used to analyze the difference in distribution of miRNAs gene polymorphisms between UC group and normal control group, as well as the effects of miRNAs gene variations on the clinicopathological characteristics and 14-week clinical response to VDZ treatment of UC patients.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed UC based on comprehensive clinical, colonoscopy, histopathological, laboratory, and radiographic examination results

Exclusion Criteria:

* rheumatoid arthritis, systemic lupus erythematosus, intestinal tuberculosis, ischemic enteritis, radiation enteritis, tumors, etc.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: There was no statistically significant difference in the gender ratio, average age, and proportion of smokers between UC group and normal control group. All study subjects are from the Zhejiang Han population who are not related by blood.
Sampling Method: Probability Sample
Enrollment: 926 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Genotypes of miRNAs | Baseline
  multiplex polymerase chain reaction-ligase detection reaction technique

CONTACTS AND LOCATIONS:
Locations (1):
- the Second Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No